CLINICAL TRIAL: NCT00544401
Title: Effect of Hypnosis and Acupuncture (Hypnopuncture) on Pregnancy Rates Following Assisted Reproductive Treatment (IVF/ICSI): A Pilot Study
Brief Title: Hypnopuncture for In Vitro Fertilization (IVF)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of participants
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Dr. Noah Samuels, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP.IVF.07
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Infertility
Keywords: infertility; in vitro fertilization; intracytoplasmic sperm implantation; acupuncture; hypnosis; hypnopuncture
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Hypnopuncture Treatment
  Interventions: Other: Hypnopuncture (Hypnosis+Acupuncture)
- 2 (No Intervention): Conventional IVF/ICSI treatment only

INTERVENTIONS:
Other: Hypnopuncture (Hypnosis+Acupuncture) — hypnosis and acupuncture
  Arms: 1

SUMMARY:
Infertility is a common and distressful problem for many couples, with assisted reproductive techniques (ART) such as IVF and ICSI, with slightly more than 34% pregnancies per cycle. Acupuncture is an ancient Chinese treatment in which thin needles are inserted into various points along the skin, harmonizing" the body's "energy. Acupuncture has been found to increase pregnancy rates following IVF/ICSI treatments, and is believed to affect ovulation and fertility through elevation of beta-endorphin release and GnRH secretion, as well as reduced sympathetic response with increased blood flow to the uterus. The sympatho-inhibitory properties and impact on beta-endorphin levels of acupuncture, as well as its efficacy in treating depression, may be helpful in reducing stress among women undergoing fertility treatments as well. Hypnosis is a mind-body technique which uses suggestions during a relaxed state to promote healing. Hypnosis can also significantly reduce the sympathetic response, and is believed to produce uterine relaxation and quiescence during embryo transfer (ET), which may lead to a reduction in embryo displacement from the uterine cavity. No research has been published on the use of hypnosis with acupuncture (hypnopuncture) in ART.

This is a pilot study to evaluate the effect of a combined regimen of hypnopuncture on clinical pregnancy rates in women undergoing IVF/ICSI following two failed cycles. During the initial pre-treatment meeting, participants who fulfill all inclusion criteria and none of the exclusion criteria will undergo hypnotic induction, followed by suggestions for increased uterine blood flow. On the day of embryo transfer, participants will be randomly divided into either treatment or no-treatment groups. Treatment will consist of the insertion of acupuncture needles into pre-determined points, to be followed by a hypnosis pre-recorded hypnosis session, as described above. Patients in the control group will receive standard care without hypnopuncture and those participants in this group who do not conceive following the 3rd cycle will be treated with hypnopuncture during the 4th cycle, following ET. A total of 100 women will be enrolled, 50 in each arm of the study.

ELIGIBILITY:
Inclusion Criteria:

* Females patients age 18 years and older
* Primary infertility with negative endocrinology and US findings on evaluation
* Following two failed cycles of either IVF or ICSI, defined as no clinical pregnancy (presence of fetal sac on ultrasound examination 6 weeks after embryo transfer).
* No underlying Axis 1 psychiatric disorder
* Ability to comply with study protocol

Exclusion Criteria:

* Patients displaying symptoms of overt Axis-1 psychopathology such as schizophrenia or severe depression.
* Current use of any CAM therapy
* Current use of any fertility treatment other than those prescribed by the fertility clinic.
* Inability to comply with the study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-11; Primary Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy - at least one intrauterine gestational sac on ultrasound scan at 3 weeks following embryo transfer | 3 weeks

SECONDARY OUTCOMES:
Implantation Rate - no. of gestational sacs/no. of transferred embryos (%) | 12 weeks
Ongoing pregnancy - viable intrauterine fetus at 12 weeks gestation | 12 weeks
Pregnancy rate following treatment of control group at 4th cycle | 12 weeks
Safety of hypnopuncture | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Noah Samuels, MD, Principal Investigator — Center for Integrative Complementary Medicine, Shaare Zedek Medical Center, Jerusalem, Israel.
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel